CLINICAL TRIAL: NCT05738824
Title: Natural History of Inflammatory Muscle Diseases
Status: Recruiting | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000894; 000894-AR
Record Dates: First submitted 2023-02-18; First posted 2023-02-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01-13

CONDITIONS: Inflammation In Skeletal Muscle
Keywords: Polymyositis; Dermatomyositis; Childhood Dermatomyositis; Natural History
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: 18 years old and up
- Patients: greater than 12 years

SUMMARY:
Objective:

To collect information and biospecimens (such as blood, muscle, and skin samples) that will be used to research causes and treatments of inflammatory muscle diseases.

Eligibility:

People aged 12 years and older with suspected or confirmed inflammatory muscle disease. Healthy volunteers aged 18 years and older are also needed.

Design:

Participants will have at least 1 clinic visit. Each visit will last 4 to 8 hours. Some may return for additional visits.

All participants will undergo these procedures (unless they are unable to):

* Physical exam, including blood and urine tests.
* Magnetic resonance imaging (MRI) scan of the thigh. Participants will lie still on a table with padding around 1 thigh. The table will slide into a tube. The scan will last for approximately 40 minutes.

Some procedures are optional:

* Muscle biopsy. An area of skin will be numbed. A quarter-inch cut will be made. Several pieces of muscle tissue, about the size of grains of rice, will be removed.
* Skin biopsy. An area of skin will be numbed. A piece of skin about a quarter inch in diameter will be removed.
* Genetic testing. Some of the samples collected may be used for genetic testing.

DETAILED DESCRIPTION:
Study Description:

This is an observational study to characterize the different types of inflammatory myopathies, understand their etiology, pathogenesis, prognosis, and response to different treatments.

Objectives:

Primary objective: Define the different types of inflammatory muscle diseases, their etiology, pathogenesis, prognostic factors, and response to different treatments.

Secondary objectives: Study different diagnostic modalities that may help to diagnose and monitor the evolution of the disease in patients with myositis.

Endpoints:

Primary endpoint: Severity of muscle, skin, pulmonary, and joint involvement. Study of the immune dysregulation, transcriptomic changes, and genetic modifications in patients with inflammatory muscle diseases.

Secondary endpoints: Utility of standard of care laboratory, radiologic, electrophysiologic, and clinical studies to diagnose and monitor the evolution of the disease in patients with myositis.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Ability of subject, or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent and/or assent document.

2a. Patients are adults and minors of age 12 or older, with possible inflammatory myopathy (suspected or confirmed)

OR

2b. Healthy volunteers will be adults aged 18 or older.

EXCLUSION CRITERIA:

1. Unwilling to participate in research studies or to provide research samples or data.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with possible inflammatory muscle disease (suspected or confirmed), and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2032-02-25 (Estimated); Study Completion 2032-02-25 (Estimated)

PRIMARY OUTCOMES:
Define the different types of inflammatory muscle diseases, their etiology, pathogenesis, prognostic factors, and response to different treatments. | End of each visit
  Severity of muscle, skin, pulmonary, and joint involvement. Study of the immune dysregulation, transcriptomic changes, and genetic modifications in patients with inflammatory muscle diseases.

SECONDARY OUTCOMES:
Study different diagnostic modalities that may help to diagnose and monitor the evolution of the disease in patients with myositis. | at baseline
  Utility of standard of care laboratory, radiologic, electrophysiologic, and clinical studies to diagnose and monitor the evolution of the disease in patients with myositis.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L Mammen, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Casal-Dominguez M, Pinal-Fernandez I, Huapaya J, Albayda J, Paik JJ, Johnson C, Silhan L, Mammen AL, Danoff SK, Christopher-Stine L. Efficacy and adverse effects of methotrexate compared with azathioprine in the antisynthetase syndrome. Clin Exp Rheumatol. 2019 Sep-Oct;37(5):858-861. Epub 2019 Apr 29. PMID 31074729
- [Background] Albayda J, Pinal-Fernandez I, Huang W, Parks C, Paik J, Casciola-Rosen L, Danoff SK, Johnson C, Christopher-Stine L, Mammen AL. Antinuclear Matrix Protein 2 Autoantibodies and Edema, Muscle Disease, and Malignancy Risk in Dermatomyositis Patients. Arthritis Care Res (Hoboken). 2017 Nov;69(11):1771-1776. doi: 10.1002/acr.23188. PMID 28085235
- [Background] Pinal-Fernandez I, Mecoli CA, Casal-Dominguez M, Pak K, Hosono Y, Huapaya J, Huang W, Albayda J, Tiniakou E, Paik JJ, Johnson C, Danoff SK, Corse AM, Christopher-Stine L, Mammen AL. More prominent muscle involvement in patients with dermatomyositis with anti-Mi2 autoantibodies. Neurology. 2019 Nov 5;93(19):e1768-e1777. doi: 10.1212/WNL.0000000000008443. Epub 2019 Oct 8. PMID 31594859
- [Background] Pinal-Fernandez I, Casal-Dominguez M, Derfoul A, Pak K, Plotz P, Miller FW, Milisenda JC, Grau-Junyent JM, Selva-O'Callaghan A, Paik J, Albayda J, Christopher-Stine L, Lloyd TE, Corse AM, Mammen AL. Identification of distinctive interferon gene signatures in different types of myositis. Neurology. 2019 Sep 17;93(12):e1193-e1204. doi: 10.1212/WNL.0000000000008128. Epub 2019 Aug 21. PMID 31434690
- [Background] Pinal-Fernandez I, Casal-Dominguez M, Derfoul A, Pak K, Miller FW, Milisenda JC, Grau-Junyent JM, Selva-O'Callaghan A, Carrion-Ribas C, Paik JJ, Albayda J, Christopher-Stine L, Lloyd TE, Corse AM, Mammen AL. Machine learning algorithms reveal unique gene expression profiles in muscle biopsies from patients with different types of myositis. Ann Rheum Dis. 2020 Sep;79(9):1234-1242. doi: 10.1136/annrheumdis-2019-216599. Epub 2020 Jun 16. PMID 32546599
- [Background] Selva-O'Callaghan A, Pinal-Fernandez I, Trallero-Araguas E, Milisenda JC, Grau-Junyent JM, Mammen AL. Classification and management of adult inflammatory myopathies. Lancet Neurol. 2018 Sep;17(9):816-828. doi: 10.1016/S1474-4422(18)30254-0. PMID 30129477
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000894-AR.html